CLINICAL TRIAL: NCT02549222
Title: A Prospective, Open Label, Post Marketing Surveillance Study Following Transfusion of INTERCEPT Platelet Components
Brief Title: A Open Label, Post Marketing Surveillance Study Following Transfusion of INTERCEPT Platelet Components
Acronym: PIPER
Status: Completed | Type: Observational
Sponsor: Cerus Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CLI 00112
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Transfusion Related Acute Lung Injury
Keywords: pathogen reduction; INTERCEPT; platelet; pulmonary; ARDS; hematology; oncology; assisted ventilation; transfusion of platelet components; hematology-oncology patients
MeSH Terms: conditions — Transfusion-Related Acute Lung Injury; Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Cohort: During the Control cohort period patients will have study data collected following transfusion with only conventional PCs for up to 21 days of transfusion support, as clinically indicated in a manner that is consistent with the local standard of care.
  Interventions: Other: Standard of Care
- INTERCEPT Cohort: During the INTERCEPT phase, patients will receive only INTERCEPT PCs and will have study data collected following transfusion for up to 21 days of transfusion support, as clinically indicated in a manner that is consistent with the local standard of care.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care

SUMMARY:
This study is a prospective, non-randomized sequential cohort, open label, multi-center, non-inferiority, Phase IV surveillance study following transfusion of INTERCEPT PCs. The patient population will be hematology-oncology patients, including those undergoing hematopoietic stem cell transplant (HSCT), expected to require one or more PC transfusions.

For each participating center, the study will start with a brief pilot run-in period with a group of at least 5 patients exposed only to conventional PCs. The purpose of this pilot run-in is to evaluate study logistics and data collection methods within each study center. Data from the pilot phase will be included in the data analysis for the treatment comparison.

After the pilot run-in period, the study will be conducted in two sequential patient cohorts: 1) the Control cohort during which study patients will receive only conventional PCs, and 2) the INTERCEPT cohort during which patients will receive only INTERCEPT PCs. Patient enrollment at each Center will be monitored to target similar numbers of patients into the Control and Test Cohorts within each center. Centers may enroll Control and Test patients in ratios that vary from 2:1 to 1:2 due to institutional requirements to move rapidly to full INTERCEPT implementation, or due to availability issues with either Test or Control components. Within each Center, patient enrollment will be stratified in four categories: (1) chemotherapy only; and by use of conditioning regimens for hematopoietic stem cell transplantation (HSCT) in (2) myeloablative conditioning, (3) non-myeloablative conditioning, and (4) reduced intensity using the Center for International Blood and Marrow Transplant Research (CIBMTR) criteria. Note time from last chemotherapy treatment to first study transfusion should be no more than 30 days. To ensure both Test and Control cohorts have a similar allocation ratio (±10% per category) among the conditioning regimen strata, enrollment caps will be set for the Test cohorts, hence no Test patients will be enrolled to a stratum once the cap for the given stratum is met. Eligible patients will be enrolled in open Test strata sequentially as long as there is sufficient Test PC inventory available. Enrollment may be delayed for the Test cohort if sufficient inventory of Test PCs is not available.

DETAILED DESCRIPTION:
The study will have a pilot run-in period and two sequential cohort groups for each center.

Pilot Run-in Period The pilot run-in period will be conducted in each center with a group of at least 5 patients exposed only to conventional PCs, who provide informed consent for data collection. The purpose of this pilot run-in is to evaluate study logistics and data collection methods within each study center. Data collection will not differ from that required in the two sequential patient cohorts. The data from the pilot phase will be included in the data analysis for the treatment comparisons.

Control and INTERCEPT Cohorts Following the run-in period, the study will be conducted in two sequential cohort periods. Informed consent for data collection without study specific treatment intervention, and under patient confidentiality, will be required for both cohorts prior to any study procedure.

During the Control cohort period, patients will have study data collected following transfusion with only conventional PCs for up to 21 days of transfusion support, as clinically indicated in a manner that is consistent with the local standard of care. During the INTERCEPT phase, patients will receive only INTERCEPT PCs under the same clinical treatment guideline. Patients will be transfused with only study PCs of the assigned treatment type (Conventional or INTERCEPT) in each cohort. Patients enrolled in the Conventional control cohort will be excluded from participating in the study in the INTERCEPT cohort.

Enrollment will be stratified by study center and type of primary disease therapy (chemotherapy only or HSCT with myeloablative, non-myeloablative, or reduced intensity conditioning).

For both cohorts, patients will be supported with study PC transfusions for a maximum of 21 days or until platelet transfusion independence. Patients are considered to have achieved platelet transfusion independence if more than 5 days elapse after exposure to a study PC transfusion. When a patient achieves platelet independence, the patient will have completed the study PC transfusion period (even if they subsequently resume another cycle of platelet support).

For the pilot phase and both cohort periods, all baseline O2 saturation values if available in the medical record should be recorded on eCRF. O2 measures associated with any form of respiratory therapy (except for room air ventilation) should be recorded with the indicated respiratory therapy for each day of therapy. If multiple measures are available in the medical record on a single day, then the worst value will be recorded.

Data collection for all participants will comprise: patient baseline disease characteristics, including primary disease, type of HSCT (auto, allo, cord blood, matched related or matched unrelated) or type of chemotherapy, and medications at study entry and during the study observation period. Patient clinical respiratory status, including, if available, a chest imaging study at baseline and O2 saturation by non-invasive pulse oximetry if available in the medical record prior to the first study transfusion in each cohort period, will also be recorded.

Within each study cohort, patients will be assessed for the primary outcome measure of assisted ventilation for a maximum of 28 days (7 days surveillance following up to of 21 days of study PC transfusion support). Patients with assisted ventilation within the defined timeframe will be further assessed for ARDS using the Berlin criteria by both the Investigator (based on diagnoses documented in the medical record) and the Pulmonary Adjudication Panel. Furthermore, AEs (including TR) will be collected from the primary medical record for 24 hours following the initiation of each study PC transfusion.; SAEs (including ARDS), CSPAEs (Grade 2 or higher AEs affecting the Respiratory System) and mortality will be collected for 7 days post each study transfusion (or until hospital discharge/discontinuation of outpatient platelet transfusion support, whichever is sooner). Investigators will assess the intensity of each AE and SAE and provide their assessment of the relationship of each AE and SAE to the study transfusion. Patients who experience the outcome of assisted ventilation, ARDS, or CSPAEs will be assessed as detailed in Assessment of Pulmonary Adverse Events in the synopsis and in Protocol Section 8.1.

For patients who achieve platelet independence before Study Day 21, AEs will be collected for 24 hours after initiating the last study platelet transfusion prior to platelet independence; the outcome of assisted ventilation, SAEs, ARDS, CSPAEs, and mortality will be collected for 7 days after the last study PC transfusion prior to platelet independence (or until hospital discharge/discontinuation of outpatient platelet transfusion support, whichever is sooner).

For patients who require more than 21 days of PC transfusion support, AEs will be recorded for up to 24 hours after the initiation of the last platelet transfusion up to and including Day 21; the outcome of assisted ventilation, SAEs, ARDS, CSPAEs, and mortality will be collected for up to a maximum of 28 days (7 days after up to 21 days of platelet transfusion support),7 days after initiating the last study transfusion within the 21-day study transfusion period (or until hospital discharge/discontinuation of outpatient platelet transfusion support, whichever is sooner). The lowest daily O2 saturation values in the medical record will be recorded on the eCRF as well.

Study-specific research personnel will review the patient medical record and record study outcomes on electronic Case Report Forms (eCRF). The intensity of AEs and SAEs will be graded according to the most recent version of the Common Terminology Criteria for Adverse Events (CTCAE) classification system. TR will also be assessed following the CDC National Healthcare Safety Network (NHSN) Biovigilance Component Hemovigilance Module Surveillance Protocol (NHSN Protocol).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a hematology-oncology disorder expected to require or requiring a transfusion of one or more PCs (time from last chemotherapy treatment to first study transfusion should be 30 days or less).
* Written signed informed consent (unless exemption of individual consent is granted by the center's IRB).

Exclusion Criteria:

* Assisted ventilation (administered by intubation or tight fitting mask with PEEP or CPAP ≥ 5 cm H2O) within 30 days prior to the first study PC transfusion. In the event that PEEP or CPAP values are unavailable for prior assisted ventilation events administered by intubation or tight fitting mask, they will be interpreted as meeting the exclusion criterion. For the purposes of this study, elective intubation of pediatric patients for the short-term protection of the airway during medical or surgical procedures does not qualify as assisted ventilation, provided that there is no parenchymal pulmonary lesion 24 hours after extubation.
* Documented allergy to psoralens

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hematology-oncology disorders, including those undergoing hematopoietic stem cell transplant (HSCT), expected to require one or more PC transfusions will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2291 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients requiring treatment-emergent assisted mechanical ventilation during the study observation period. | Up to 28 days
  For the purposes of this study, assisted mechanical ventilation defined as assisted ventilation started after the initiation of the first study PC and can be administered either by intubation or tight fitting mask with positive end-expiratory pressure (PEEP) or continuous positive airway pressure (CPAP or BiPAP) ≥ 5 cm H2O, if PEEP or CPAP information is available. Assisted mechanical ventilation is selected as the primary outcome as it provides an objective measure of severe, clinically significant pulmonary injury. Patients will be assessed for the initiation of assisted ventilation within 7 days after each study PC transfusion.

SECONDARY OUTCOMES:
Time from first study PC transfusion to onset of treatment-emergent assisted mechanical ventilation. | Up to 28 days
  Time from first study Platelet Component transfusion to onset of treatment-emergent assisted mechanical ventilation.
AEs occurring within 24 hours after the initiation of a study PC transfusion | Up to 22 days
  Adverse Events occurring within 24 hours after the initiation of a study PC transfusion.
TR occurring within 24 hours after the initiation of a study PC transfusion. | Up to 22 days
  Transfusion Reactions occurring within 24 hours after the initiation of a study PC transfusion.
SAEs occurring within 7 days after each study PC transfusion | Up to 28 days
  Serious Adverse Events occurring within 7 days after each study PC transfusion
ARDS occurring within 7 days after each study PC transfusion | Up to 28 days
  Acute Respiratory Distress Syndrome occurring within 7 days after each study PC transfusion
CSPAEs occurring within 7 days after each study PC transfusion | Up to 28 days
  Clinically Serious Pulmonary Adverse Events occurring within 7 days after each study PC transfusion
Mortality within 7 days after the last study PC transfusion, or until hospital discharge/discontinuation of outpatient platelet transfusion support, whichever is sooner (all deaths and deaths due to ARDS). | Up to 28 days
  Mortality within 7 days after the last study PC transfusion, or until hospital discharge/discontinuation of outpatient platelet transfusion support, whichever is sooner (all deaths and deaths due to ARDS).

CONTACTS AND LOCATIONS:
Overall Officials: Edward L Snyder, MD, Principal Investigator — Yale New Haven Hospital
Locations (15):
- United States (15):
  - UCLA Medical Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - University of Maryland, Baltimore, Maryland
  - Beth Israel, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering, New York, New York
  - Strong Memorial Hospital, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University Hospital, Greenville, North Carolina
  - TriHealth Cancer Institute, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Derived] Wheeler AP, Snyder EL, Refaai M, Cohn CS, Poisson J, Fontaine M, Sehl M, Nooka AK, Uhl L, Spinella PC, Fenelus M, Liles D, Coyle T, Becker J, Jeng M, Gehrie EA, Spencer BR, Young P, Johnson A, O'Brien JJ, Schiller GJ, Roback JD, Malynn E, Jackups R, Avecilla ST, Liu K, Bentow S, Varrone J, Benjamin RJ, Corash LM. Acute pulmonary injury in hematology patients supported with pathogen-reduced and conventional platelet components. Blood Adv. 2024 May 14;8(9):2290-2299. doi: 10.1182/bloodadvances.2023012425. PMID 38447116
- [Derived] Delaney M, Karam O, Lieberman L, Steffen K, Muszynski JA, Goel R, Bateman ST, Parker RI, Nellis ME, Remy KE; Pediatric Critical Care Transfusion and Anemia EXpertise Initiative-Control/Avoidance of Bleeding (TAXI-CAB), in collaboration with the Pediatric Critical Care Blood Research Network (BloodNet), and the Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. What Laboratory Tests and Physiologic Triggers Should Guide the Decision to Administer a Platelet or Plasma Transfusion in Critically Ill Children and What Product Attributes Are Optimal to Guide Specific Product Selection? From the Transfusion and Anemia EXpertise Initiative-Control/Avoidance of Bleeding. Pediatr Crit Care Med. 2022 Jan 1;23(13 Suppl 1 1S):e1-e13. doi: 10.1097/PCC.0000000000002854. PMID 34989701